CLINICAL TRIAL: NCT05344885
Title: Examining the Impact of Intervention Design in Digital Parent Training for Child's Disruptive Behaviors: A Pilot Randomized Trial
Brief Title: A Pilot Trial Examining Digital Parent Training Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Amit Baumel, Senior Lecturer, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2836
Record Dates: First submitted 2022-04-07; First posted 2022-04-25 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Child Behavior Problem; Parenting; Engagement, Patient
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPT-standard (Active Comparator): A standard digital parent training intervention
  Interventions: Behavioral: DPT-Standard
- DPT-Enhanced (Experimental): Enhanced digital parent training intervention
  Interventions: Behavioral: DPT-Enhanced

INTERVENTIONS:
Behavioral: DPT-Standard — The parent training intervention includes 7 modules, recommended to be completed within 7- to 10-weeks period. Module's content includes videos and texts guiding the parent through the training process; interactive features, such as multiple-choice questions with direct feedback. Additional features embedded within the platform include downloadable materials, and a Q&A section that contains frequently asked questions.
  Arms: DPT-standard
Behavioral: DPT-Enhanced — DPT-Enhanced will include all the ingredients of DPT-Standard, but with additional features. The program itself is based on pre-defined decision rules that are either event or time based based on evidence based practice in promoting effective parental engagement. Each component includes a short learning phase, followed by a 1-2 week focusing phase. The focusing phase is designed to encourage and help parents to practice and acquire learned skills in their day-to-day lives, by making these skills more salient in their mind.
  Arms: DPT-Enhanced

SUMMARY:
The purpose of this pilot study is to preliminary examine the impact of a design mechanism aimed at increasing engagement in an unguided digital parent training program for child's behavior problems. Parents will be enrolled into one of two digital parent training intervention arms, dedifferentiated by their level of correspondence with the related deign mechanism.

DETAILED DESCRIPTION:
The purpose of this pilot study is to preliminary examine the impact of a design mechanism aimed at increasing engagement in an unguided digital parent training program for child's behavior problems. The design mechanism manipulated in this pilot relates to the extent to which program design promotes a positive behavior change. To achieve these goal two unguided digital parent training interventions, differentiated by their level of design (DPT-Standard vs. DPT-Enhanced), will be tested. This pilot aims to recruit 40-60 parents who report behavior problems in their children who will randomly receive one of the two interventions for 10 weeks.

The impact of DPT-E on user engagement and reported child behavior problems will be assessed based on comparison with DPT-Standard. Parental behaviors and sense of competence will be collected to assess the impact of intervention design on these mechanisms of change. In addition, the role of parents' motivation, and their ability to invest effort in making changes during the intervention will be assessed, to examine whether these variables moderate the impact of intervention's design on the aforementioned relationships. The investigators also aim to explore whether the relationship between usage and clinical outcomes is stronger in those using DPT-E compared with DPT-Standard.

ELIGIBILITY:
Inclusion Criteria:

1. Parents report they have a child between the ages of 3 and 7, who:
2. Has externalized behavior problems based on A) Parents report at least 1 of the two first criteria of behavior problems to be above 4 (the middle point) & the average of all items ≥ 4, on a screening scale that consists of 9 items (on a Likert scale between 1 and 7) that is based on DSM-V symptoms for ODD.

   B) Parents report ECBI Problems to be above 14 OR Intensity to be above 130.
3. Parents have access to computer at home with an Internet connection and a smartphone with a mobile data plan.
4. Parents can read and understand Hebrew.

Exclusion Criteria:

1. Parents report that the relevant child has been diagnosed with developmental delay, intellectual disability and/or autism spectrum disorder.
2. Parent and/or child are already receiving therapeutic intervention (for the child) in other setting.
3. The relevant child is treated with psychiatric medication.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Eyberg Child Behavior Inventory (ECBI) at 10 weeks | 10 weeks
  The ECBI specifies 36 behaviors commonly reported by parents of children with behavior problems. For each behavior the parent specifies how often this problem occurs on a 1-7 Likert scale (1=never; 7=always; higher scores mean worse outcome), and whether this behavior is currently a problem (0=no; 1=yes; higher scores mean worse outcome).

SECONDARY OUTCOMES:
change from Baseline Behavior and Feelings Survey Externalizing Problems at 10 weeks | 10 weeks
  The Behavior and Feelings Survey (BFS) parent report of Externalizing Problems in children and adolescents is based on summing 6 items that measure children's behavior problems on a 0-4 scale (0=not a problem; 4=a very big problem).
change from Baseline Parenting Scale (PS) at 10 weeks | 10 weeks
  Two sub-scales of the Parenting Scale, Over-reactivity (11 items) and Laxness (10 items) will be used in this study. The parent is requested to mark his typical response on a 7-point Likert scale (1-7), when 7 indicates the ineffective spectrum (higher scores mean worse outcome), and 1 indicates the effective spectrum.
change from Baseline Alabama Parenting Questionnaire (APQ) positive parenting practices at 10 weeks | 10 weeks
  3 items, 1 sub-scale: measuring positive parenting practices. Parents will be asked to mark the frequency they use each parental practice on a 5-point scale ranging from 1 (never) to 5 (always; higher scores mean better outcome).
change from Baseline Me as a Parent (MAAP) self-efficacy at 10 weeks | 10 weeks
  4 items, 1 sub-scale measures general parental self-efficacy. Responses range on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree (higher scores mean better outcome).
change from Baseline Parenting Tasks Checklist (PTC) self-efficacy at 10 weeks | 10 weeks
  12 items, 2 sub-scales: behavioral self-efficacy (6 items), setting self-efficacy (6 items). Parents are asked to rate each item on a scale ranges from 0 to 100 (0=Certain I can't do it, 100=Certain I can do it; higher scores mean better outcome).
Program Usage Time | through program completion, an average of 10 weeks
  Time on the platform (measured in minutes)
Program Logins | through program completion, an average of 10 weeks
  Number of user logins to the platform
Number of Modules completed | through program completion, an average of 10 weeks
  The number of program Modules that were completed while using the program

CONTACTS AND LOCATIONS:
Overall Officials: Amit Baumel, PhD, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No